CLINICAL TRIAL: NCT02066363
Title: Best Nutritional Care in Cancer Patients. A Comparative Randomized Study of Supplemental Parenteral Nutrition to Patients With GI Cancer Compared to Best Supportive Nutritional Care
Brief Title: Study of Parenteral Nutrition to Patients With Gastrointestinal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment very time consuming, too few wanting participation
Sponsor: Odense University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Region of Southern Denmark (Other); Danish Cancer Society (Other); Aase and Ejnar Danielsens Foundation (Other); Hartmann Fonden (Other); Knud and Edith Eriksen Memorial Fund (Unknown); Merchant M. Brogaard and Wife Memorial fund (Unknown); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Sine Obling, MD, Registrar, ph.d student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HPN 01
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Gastrointestinal Cancer; Dietary Modification; Cancer Cachexia; Quality of Life; Body Composition, Beneficial
Keywords: Bioelectrical impedance; Parenteral nutrition; Malnutrition; Quality of life.; Cancer cachexia; Body composition
MeSH Terms: conditions — Gastrointestinal Neoplasms; Glucocorticoid Receptor Deficiency; Hyperphagia; Malnutrition | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Best nutritional Care (Active Comparator): Best supportive nutritional care and dietician advise
  Interventions: Dietary Supplement: Dietician advise
- Parenteral nutrition (Experimental): Supplemental Parenteral Nutrition and dietician advise. Supplemental parenteral Nutrition 30% of estimated needs. Parenteral nutrition given at home, administered by a nurse. The patient will be seen at the Outpatient Clinic every 6th week, talk to dietician and a doctor.
  Interventions: Dietary Supplement: Dietician advise; Dietary Supplement: Parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Dietician advise — Dietician advise 5 times, during 24weeks. Prescription of a diet plan if wanted from the patient.
  Other Names: Best supportive Nutritional care,
Dietary Supplement: Parenteral nutrition — Supportive parenteral nutrition.
  Arms: Parenteral nutrition

SUMMARY:
Clinical background: Weight loss is a common problem in patients suffering from gastrointestinal cancer. It is demonstrated that the prognosis for cancer patients with weight loss is worse than that for weight stable patients. Malnutrition in cancer patients is associated with a poor prognosis and is an important predictor of mortality. Supplementation with home parenteral nutrition in aphagic and terminal patients has shown improved quality of life, energy balance, body composition and prolonged survival.

Aim: The aim of this study is primarily to study the effects of supplementation with parenteral nutrition, to patients with advanced incurable gastrointestinal cancer on lean body-mass and body composition. Patients found to be at nutritional risk will be included in the study and will be randomized to either best supportive nutritional care or best supportive nutritional care and supplemental Parenteral Nutrition.

Design: This study is a controlled, randomized trial with two parallel study arms. The study will include patients with advanced GI cancers at nutritional risk, performance status 0-2 and with an expected survival of a minimum of 3 months.

A total of 100 patients are planned to be enrolled and randomized to either best supportive nutritional care or best supportive nutritional care and supplemental parenteral Nutrition.

Primary endpoint is improvement of lean body mass, and by that improvement of quality of life, performance status and cancer treatment tolerance.

Discussion: The planned study will provide important information about the effect of parenteral nutrition in a patient group with advanced gastrointestinal cancer. Palliative treatment strategies are set up to improve quality of life as well as prolongation of life. Parenteral nutrition in this patient group may indeed contribute to both these aspects of palliation.

DETAILED DESCRIPTION:
Randomizing. The patients will be enrolled in the study, by block randomizing using a computer generated list, stratifying in respect to performance status 0 and 1 in opposite to PS 2 for the first 10 patients enrolled in the study.

To make the two treatment groups comparable, the patients number 11-100 enrolled in the study will be placed in the treatment groups using the minimization method. Using the minimization method the prognostic factors for age, diagnosis and performance status at the enrollment, will be considered to make the treatment groups similar.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-resectable GI-Cancer
* at nutritional risk; having lost 5% of body weight during the previous 3 months or has failed to reach intake by 25% in the last 2 weeks.
* At performance status 0-2
* Life expectancy more than 3 months.
* Age over 18 years old.
* Able to give written consent

Exclusion Criteria:

* Gastrointestinal obstruction or failure.
* Immune deficiency diseases (apart from the cancer disease. )
* Current infection or sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-03-01; Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | Six months
  Measured by using bioelectrical impedance analysis.

SECONDARY OUTCOMES:
Time to to exacerbate Quality of Life | six months
  Assessment of quality of life by European Organization for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ30)

OTHER OUTCOMES:
frequency of readmission to the Hospital | 6 months
  Number of admissions
Survival in study | 6 months
  Time to event; survival time in study

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kjeldsen, ph.d, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Obling SR, Wilson BV, Pfeiffer P, Kjeldsen J. Home parenteral nutrition increases fat free mass in patients with incurable gastrointestinal cancer. Results of a randomized controlled trial. Clin Nutr. 2019 Feb;38(1):182-190. doi: 10.1016/j.clnu.2017.12.011. Epub 2017 Dec 21. PMID 29305245